CLINICAL TRIAL: NCT04919382
Title: A Randomized, Multi-Cohort Phase II Trial of Temozolomide and Atezolizumab for Subsequent Line Treatment for Small Cell Lung Cancer
Brief Title: Temozolomide and Atezolizumab for Subsequent Line for the Treatment of Metastatic or Recurrent Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dwight Owen (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Dwight Owen, Sponsor Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC LUN20-462; NCI-2021-05580 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Extensive Stage Lung Small Cell Carcinoma; Metastatic Lung Small Cell Carcinoma; Recurrent Lung Small Cell Carcinoma; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Small Cell Lung Carcinoma; Lung Neoplasms | interventions — atezolizumab; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cohort I (atezolizumab, temozolomide) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on day 1 and temozolomide PO QD on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Atezolizumab; Drug: Temozolomide
- Cohort II (atezolizumab, temozolomide) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on day 1. Patients also receive temozolomide PO QD on days 1-14 of cycle 1 and days 1-21 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Atezolizumab; Drug: Temozolomide

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase II trial studies the effects of temozolomide and atezolizumab as second or third line treatment for patients with small cell lung cancer that has spread to other places in the body (metastatic) or has come back (recurrent). Chemotherapy drugs, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving temozolomide and atezolizumab as second or third line treatment may help prolong survival in patients with small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To estimate the efficacy of atezolizumab and temozolomide in two dosing schedules for patients with metastatic small-cell lung cancer (SCLC) who progress after chemoimmunotherapy.

SECONDARY OBJECTIVES:

I. To evaluate the safety profile and toxicity of combination atezolizumab and temozolomide in two dosing schedules as per Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

II. To evaluate the progression free survival (PFS) and overall survival (OS) of patients treated with combination atezolizumab and temozolomide.

III. To evaluate the intracranial PFS rate at 6 months (icPFS6) of patients with SCLC treated with atezolizumab and temozolomide.

CORRELATIVE/EXPLORATORY OBJECTIVES:

I. Explore association of myeloid-derived suppressor cell (MDSC) levels at baseline biomarker status from tumor biopsy samples and peripheral blood and correlate these with clinical parameters (including overall response rate [ORR], OS and toxicity).

II. To evaluate changes in MDSC induced by different dosing of temozolomide. III. To explore post-translational modifications of PD-L1 by mass spectrometry.

OUTLINE: Patients are randomized to 1 of 2 cohorts.

COHORT I: Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1 and temozolomide orally (PO) once daily (QD) on days 1-5. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients receive atezolizumab IV over 30-60 minutes on day 1. Patients also receive temozolomide PO QD on days 1-14 of cycle 1 and days 1-21 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization for release of personal health information

  * NOTE: HIPAA authorization may be included in the informed consent or obtained separately
* Age >= 18 years at the time of consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2 within 28 days prior to registration
* Have histologically or cytologically-documented diagnosis of extensive stage (i.e. metastatic and/or recurrent) small cell lung cancer and have progressed or recurred after platinum-based chemotherapy with immunotherapy. Eligible patients will be defined as follows:

  * "Sensitive" Disease: Patients who had one previous line of chemotherapy and relapsed after > 90 days of completion of treatment
  * "Resistant" Disease: Patients with no response to first-line chemo-immunotherapy or progression < 90 days after completing treatment
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 within 28 days prior to registration
* Maximum of 3 prior lines of systemic therapy is allowed in the setting of metastatic disease. Patients who recur after treatment for limited state disease, and who receive first line metastatic treatment with chemo-immunotherapy would be considered eligible upon progression on chemo-IO in the metastatic setting
* Absolute neutrophil count (ANC) >= 1.5 K/mm^3 (obtained within 28 days prior to registration)
* Platelets >= 100,000 / mcL (obtained within 28 days prior to registration)
* Serum creatinine =< 2.0 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 50 mL/min as estimated by Cockcroft and Gault formula for subject with creatinine levels > 2 x institutional ULN (obtained within 28 days prior to registration)
* Bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN

  * Patients with known Gilbert disease: serum bilirubin =< 3 x ULN) (obtained within 28 days prior to registration)
* Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) =< 3 X ULN OR =< 5 X ULN for subjects with liver metastases (obtained within 28 days prior to registration)
* Albumin > 2.5 g/dL (obtained within 28 days prior to registration)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN for patients not receiving therapeutic anticoagulation (obtained within 28 days prior to registration)

  * For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN for patients not receiving therapeutic anticoagulation (obtained within 28 days prior to registration)

  * For patients receiving therapeutic anticoagulation: stable anticoagulant regimen
* Females of childbearing potential must have a negative serum or urine pregnancy test within 14 days prior to registration
* For women of childbearing potential: agreement to remain abstinent (refrain from vaginal intercourse) or use contraceptive methods and agreement to refrain from donating eggs, as defined below:

  * Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 5 months after the final dose of atezolizumab or temozolomide. Women must refrain from donating eggs during this same period
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone releasing intrauterine devices, and copper intrauterine devices
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, sympto-thermal, or post ovulation methods) and withdrawal are not adequate methods of contraception
* For men able to father a child: agreement to remain abstinent (refrain from vaginal intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

  * With a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 3 months after the final dose of temozolomide to avoid exposing the embryo. Men must refrain from donating sperm during this same period
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study
* Availability of archival tissue, preferably a recent formalin-fixed, paraffin-embedded (FFPE) tumor tissue block. A recently obtained archival FFPE tumor tissue block from a primary or metastatic tumor resection or biopsy can be provided if it was obtained within 1 year of trial screening. Patients with tumor specimens older than 1 year, or who do not have biopsy specimen may still be eligible if deemed so by the sponsor-investigator.
* Be willing to provide peripheral blood samples at specified time-points during the study
* Life expectancy greater than 3 months as determined by the enrolling physician or protocol designee
* Ability to swallow and retain oral medication

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has received prior temozolomide therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are not eligible for this trial
* Symptomatic central nervous system (CNS) metastases or untreated or actively progressing CNS metastases. Subjects with asymptomatic CNS metastases (treated or untreated) will be eligible provided all of the following criteria are met.

  1. Measurable disease, per RECIST v1.1, must be present outside the CNS.
  2. The patient has no history of intracranial hemorrhage or spinal cord hemorrhage.
  3. The patient has not undergone stereotactic radiotherapy within 7 days prior to initiation of study treatment, whole-brain radiotherapy within 14 days prior to initiation of study treatment, or neurosurgical resection within 28 days prior to initiation of study treatment.
  4. The patient has no ongoing requirement for corticosteroids as therapy for CNS disease at the time of study treatment.
  5. If the patient is receiving anti-convulsant therapy, the dose is considered stable and appropriate by the treating physician.
  6. Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla, or spinal cord).

     * NOTE: Subjects who are symptomatic and have not undergone prior brain imaging must undergo a head computed tomography (CT) scan or brain MRI within 28 days prior to registration to exclude brain metastases
     * NOTE: A subject with previously treated brain metastasis may be considered if they have completed their treatment for brain metastasis at least 2 weeks prior to study registration and all of the above criteria are met.
* Clinically significant acute infection requiring systemic antibacterial, antifungal, or antiviral therapy including:

  * Tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and TB testing in line with local practice)
  * Hepatitis B (known positive HBV surface antigen [HBsAg] result)
  * Hepatitis C, or
  * Human immunodeficiency virus (positive HIV 1/2 antibodies)
  * NOTES: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. In patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA). Subjects with HIV/acquired immunodeficiency syndrome (AIDS) with adequate antiviral therapy to control viral load (i.e undetectable) would be allowed if they are stable and have been on treatment for >= 4 weeks prior to first dose of study drug(s). Subjects with viral hepatitis with controlled viral load would be allowed while on suppressive antiviral therapy. Testing not required
* Has had prior chemotherapy, immunotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with =< grade 2 neuropathy or alopecia due to chemotherapy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
  * Note: Subjects with irreversible toxicity that in the opinion of the treating physician is not reasonably expected to be exacerbated by the investigational product may be included (e.g., hearing loss, hormone deficiency requiring replacement therapy)
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions:

  * Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
  * Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover =< 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (more than once monthly). Patients with indwelling catheters (e.g., PleurX) are allowed.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium >12 mg/dL or corrected serum calcium > ULN)
* History of leptomeningeal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-01-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Investigator-assessed objective response rate (ORR) | Up to 2 years
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Response will be defined by a confirmed complete response (CR) or confirmed partial response (PR). Response will be defined for patients with measurable disease and who receive at least one dose of combination treatment. ORR rate will be calculated as the proportion of patients with RECIST-based PR or CR divided by the total number of evaluable patients. Exact binomial 90% and 95% confidence intervals for the true PR+CR response rate will be calculated.

SECONDARY OUTCOMES:
Treatment related adverse events | Up to 2 years
  Defined by the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.
Progression free survival (PFS) | From initiation of investigational therapy until the criteria for disease progression is met as defined by RECIST1.1 or death as a result of any cause, assessed up to 2 years
  Will be estimated with Kaplan-Meier method. Median with 95% confidence interval will be calculated.
Intracranial PFS | At 6 months from start of investigational therapy
  Defined as the percentage of patients without intracranial disease progression (including patients with and without intracranial disease at baseline), including development of new lesions, development of symptomatic lesions or leptomeningeal disease, or intervention required for disease control (such as radiation or surgery). Will be estimated with Kaplan-Meier method. Median with 95% confidence interval will be calculated.
Overall survival | Date of initiation of investigational therapy to date of death from any cause, assessed up to 2 years
  Will be estimated with Kaplan-Meier method. Median with 95% confidence interval will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Dwight Owen, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (5):
- United States (5):
  - University of Illinois Cancer Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Wisconsin, Madison, Wisconsin